CLINICAL TRIAL: NCT06654986
Title: The Importance of Amino Acid Availability in Modulating the Muscle Anabolic Response to β2-adrenergic Stimulation.
Brief Title: Muscle Anabolic Response to β2-adrenergic Stimulation With Increased Amino Acid Availability.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SALM_chron
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Beta2-adrenergic stimulation; Amino acid availability; Skeletal muscle hypertophy
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Intervention Model Description: Thirty-six healthy, well-trained men and women will be randomized into three distinct groups, each receiving one of the following interventions: 1) salmeterol with amino acid availability, 2) salmeterol, or 3) a placebo, administered twice daily over a 6-week intervention period. This design aims to elucidate the impact of amino acid availability on the muscle anabolic response to beta2-adrenergic stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Salmeterol + amino acid availability (Experimental): The participants will be administered salmeterol from an inhaler device and amino acid availability (protein powder in a shaker) daily during a 6-week intervention.
  Interventions: Drug: Salmeterol + amino acid availability
- Salmeterol + placebo (Experimental): The participants will be administered salmeterol from an inhaler device. Furthermore they will be administered placebo (carbo fuel in a shaker) daily during a 6-week intervention.
- Placebo + placebo (Placebo Comparator): The participants will be administered placebo from an inhaler device. Furthermore they will be administered placebo (carbo fuel in a shaker) daily during a 6-week intervention.
  Interventions: Drug: Placebo + placebo

INTERVENTIONS:
Drug: Salmeterol + amino acid availability — The participants will be administered 200 µg salmeterol (8 puffs) from a MDI device and 40 g amino acid availability (clear whey in a shaker with water) daily during a 6-week intervention. Participants will be instructed to provide documentation of both the inhalation and the shaker intake via video.
  Arms: Salmeterol + amino acid availability
Drug: Salmeterol + placebo — The participants will be administered 200 µg salmeterol (8 puffs) from a MDI device. Furthermore they will be administered 80 g placebo (carbo fuel in a shaker with water) daily during a 6-week intervention. Participants will be instructed to provide documentation of both the inhalation and the shaker intake via video.
Drug: Placebo + placebo — The participants will be administered placebo (8 puffs) from a MDI device. Furthermore they will be administered 80 g placebo (carbo fuel in a shaker with water) daily during a 6-week intervention. Participants will be instructed to provide documentation of both the inhalation and the shaker intake via video.
  Arms: Placebo + placebo

SUMMARY:
The purpose of the project is to investigate the effect of amino acid availability on the muscle anabolic response to beta2-adrenergic stimulation in young healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Physically active >5 hours a week
* Maximum oxygen uptake classified as high or very high

Exclusion Criteria:

* Active smoker currently or within the past 5 years
* Regular intake of medication deemed by the responsible study physician to affect the test parameters (hormonal contraception is accepted for women)
* Chronic or acute illness deemed by the responsible study physician to affect the test parameters
* Deviation from the study protocol
* Lean mass index >21 kg/m²
* Pregnancy
* Smoker
* Blood donation during the past 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle hypertrophy | Through study completion, an average on 7 weeks
  Muscle hypertrophy measured using Dual-energy X-ray Absorptiometry (DXA).

SECONDARY OUTCOMES:
Quadriceps strength | Through study completion, an average on 7 weeks
  Maksimal torque (Nm) achieved during isometric contraction
Power output during sprint testing | Through study completion, an average on 7 weeks
  Power output measured in Watts during a sprint on a bike ergometer
Power output during time trial | Through study completion, an average on 7 weeks
  Mean power output measured in Watts during a time trial on a bike ergometer

OTHER OUTCOMES:
Maximal oxygen uptake | Through study completion, an average on 7 weeks
  Maximal oxygen uptake measured during an incremental test to exhaustion on a bike ergometer.

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided